CLINICAL TRIAL: NCT02186873
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, an Anti-TNFα Monoclonal Antibody, Administered Intravenously, in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study of Golimumab in Participants With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103795; CNTO148AKS3001 (Other: Janssen Research & Development, LLC); 2014-000241-74 (EudraCT Number)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Golimumab; SIMPONI
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Treatment Group 1: Placebo then Golimumab (Experimental): Participants will receive intravenous infusions of placebo at Weeks 0, 4 and 12. At Week 16, all participants receiving placebo will begin receiving intravenous infusions of golimumab 2 milligram per kilogram (mg/kg) at Weeks 16, 20 and thereafter every 8 weeks up to Week 52.
  Interventions: Drug: Placebo; Drug: Golimumab
- Treatment Group 2: Golimumab (Experimental): Participants will receive intravenous infusions of golimumab 2 mg/kg at Weeks 0, 4 and thereafter every 8 weeks up to Week 52. At Week 16, participants will receive a placebo infusion to maintain the blind.
  Interventions: Drug: Placebo; Drug: Golimumab

INTERVENTIONS:
Drug: Placebo — Participants will receive matching placebo.
Drug: Golimumab — Participants will receive 2mg/kg of intravenous infusions of golimumab .

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravenously (administration of a fluid into the vein) administered golimumab 2 milligram per kilogram (mg/kg) in participants with active ankylosing spondylitis (chronic inflammatory disease of unknown etiology that involves the sacroiliac joints, and often the axial skeleton, entheses, and peripheral joints).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study drug assigned by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study of golimumab compared with placebo in participants with active ankylosing spondylitis. The study comprises of 4 phases: Screening phase (up to 6 weeks), Double-blind placebo-controlled phase (Week 0 to Week 16), Active treatment phase (Week 16 to Week 52), and Safety follow-up phase (8 weeks from last study drug administration). Total duration of the study will be 60 weeks per participant. Eligible Participants will be randomly assigned to either Treatment group 1: Placebo or Treatment group 2: Golimumab. Participants randomized to Placebo group, will receive intravenous infusions of placebo at Weeks 0, 4 and 12. At Week 16, all participants receiving placebo will begin receiving intravenous infusions of golimumab (2 mg/kg) at Weeks 16, 20 and thereafter every 8 weeks up to Week 52. Participants randomized to Golimumab group, will receive intravenous infusions of golimumab 2 mg/kg at Weeks 0, 4 and thereafter every 8 weeks up to Week 52. At Week 16, participants randomized to golimumab group will receive a placebo infusion to maintain the blind. The efficacy will be assessed primarily by measuring percentage of participants who achieve a 20 percent improvement from baseline in the assessment in ankylosing spondylitis (ASAS) at Week 16. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of definite ankylosing spondylitis for at least 3 months based on modified New York radiographic and clinical criteria
* Participants with symptoms of active disease at screening and at baseline
* Participant has either an inadequate response to at least 2 non-steroidal anti-inflammatory drugs (NSAID) over a 4 week period in total with maximal recommended doses of NSAIDs, or is unable to receive a full 4 weeks of maximal NSAID therapy because of intolerance, toxicity, or contraindications to NSAIDs
* Participants with C- reactive protein (CRP) level of greater than or equal to (>=) 0.3 milligram per deciliter (mg/dL) at screening
* Additional protocol-defined inclusion criteria apply

Exclusion Criteria:

* Participant with other inflammatory diseases that might confound the evaluations of benefit from the golimumab therapy
* Pregnant or lactating females
* Participants with chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection, including tuberculosis
* Participants who had a serious infection (including but not limited to, hepatitis, pneumonia, sepsis, or pyelonephritis), or have been hospitalized for an infection, or have been treated with intravenous (IV) antibiotics for an infection within 2 months prior to first administration of study agent
* Additional protocol-defined exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (45):
- United States (11):
  - Glendale, Arizona
  - Mesa, Arizona
  - La Palma, California
  - Granger, Indiana
  - St Louis, Missouri
  - Orchard Park, New York
  - Salisbury, North Carolina
  - Middleburg Heights, Ohio
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Houston, Texas
- Maroochydore, Australia
- Canada (3):
  - St. John's, Newfoundland and Labrador
  - Burlington
  - Trois-Rivières
- Germany (7):
  - Bad Doberan
  - Berlin
  - Erfurt
  - Hamburg
  - Planegg
  - Ratingen
  - Zerbst
- Chihuahua City, Mexico
- Poland (6):
  - Bydgoszcz
  - Bytom
  - Nadarzyn
  - Nowa Sól
  - Poznan
  - Warsaw
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tver'
- South Korea (5):
  - Ansan
  - Daegu
  - Gwangju
  - Seongdong-Gu
  - Seoul
- Ukraine (6):
  - Chernihiv
  - Dnipropetrovsk
  - Kyiv
  - Odesa
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] Deodhar A, Shiff NJ, Gong C, Chan EKH, Hsia EC, Lo KH, Akawung A, Kim L, Xu S, Reveille JD. Effect of Intravenous Golimumab on Fatigue and the Relationship with Clinical Response in Adults with Active Ankylosing Spondylitis in the Phase 3 GO-ALIVE Study. Rheumatol Ther. 2023 Aug;10(4):983-999. doi: 10.1007/s40744-023-00556-y. Epub 2023 Jun 15. PMID 37322274
- [Derived] Deodhar AA, Shiff NJ, Gong C, Hsia EC, Lo KH, Kim L, Xu S, Reveille JD. Efficacy and Safety of Intravenous Golimumab in Ankylosing Spondylitis Patients With Early and Late Disease Through One Year of the GO-ALIVE Study. J Clin Rheumatol. 2022 Aug 1;28(5):270-277. doi: 10.1097/RHU.0000000000001853. Epub 2022 Jun 1. PMID 35653615
- [Derived] Husni ME, Deodhar A, Schwartzman S, Chakravarty SD, Hsia EC, Leu JH, Zhou Y, Lo KH, Kavanaugh A. Pooled safety results across phase 3 randomized trials of intravenous golimumab in rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. Arthritis Res Ther. 2022 Mar 21;24(1):73. doi: 10.1186/s13075-022-02753-6. PMID 35313978
- [Derived] Reveille JD, Hwang MC, Danve A, Kafka S, Peterson S, Lo KH, Kim L, Hsia EC, Chan EKH, Deodhar A. The effect of intravenous golimumab on health-related quality of life and work productivity in adult patients with active ankylosing spondylitis: results of the phase 3 GO-ALIVE trial. Clin Rheumatol. 2021 Apr;40(4):1331-1341. doi: 10.1007/s10067-020-05342-7. Epub 2020 Sep 14. PMID 32926247
- [Derived] Deodhar A, Reveille JD, Harrison DD, Kim L, Lo KH, Leu JH, Hsia EC. Safety and Efficacy of Golimumab Administered Intravenously in Adults with Ankylosing Spondylitis: Results through Week 28 of the GO-ALIVE Study. J Rheumatol. 2018 Mar;45(3):341-348. doi: 10.3899/jrheum.170487. Epub 2017 Dec 15. PMID 29247154

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 312 participants screened, 208 participants were randomized (105 to golimumab 2 milligram per kilogram [mg/kg] and 103 to placebo group) and treated.
Groups:
- Group 1: Placebo Then Golimumab: Participants received placebo intravenous (IV) infusions at Weeks 0, 4, and 12. At Week 16 participants were crossed over to golimumab and received IV golimumab 2 mg/kg infusions at Weeks 16, 20, and every 8 weeks (q8w) thereafter through Week 52.
- Group 2: Golimumab: Participants received IV golimumab 2 mg/kg infusion at Weeks 0, 4 and then q8w thereafter through Week 52. Participants received a placebo infusion at Week 16 to maintain the treatment blind.
Period: Overall Study
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Started | 103 | 105
End of Control Period | 99 (Participants taking placebo crossed over to golimumab) | 105 (Participants continued to receive golimumab)
Completed | 94 | 97
Not Completed | 9 | 8
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 105 | 207
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (10.75) | 38.4 (10.11) | 38.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 77 | 86 | 163
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2
  Germany | 3 | 5 | 8
  Mexico | 3 | 3 | 6
  Poland | 38 | 30 | 68
  Russian Federation | 16 | 14 | 30
  South Korea | 8 | 10 | 18
  Ukraine | 25 | 34 | 59
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieved at Least 40 Percent Improvement From Baseline in the Assessment of SpondyloArthritis International Society (ASAS 40) at Week 16
Description: An ASAS 40 response is defined as >=40% improvement from baseline in 3 of 4 domains: patient's global assessment of disease activity (0=very well, 10=very poor), total back pain (0=no pain, 10=most severe pain), function (self-assessment using BASFI (0=no functional impairment to 10=maximal impairment), inflammation (0=none, 10=very severe) with an absolute improvement of at least 2 (0-10 cm VAS), and no deterioration in the remaining domain.
Time Frame: Week 16
Population: FAS included all participants who were randomized in the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 103 | 105
Percentage of Participants | 8.7 | 47.6

2. Secondary Outcome: Percentage of Participants Who Achieved at Least 50 Percent Improvement From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 16
Description: The BASDAI is a self-assessment tool to determine disease activity using a VAS of 0-10 cm (0=none and 10=very severe) participant's answered 6 questions measuring fatigue, spinal pain, joint pain, enthesitis, and morning stiffness. The final BASDAI is calculated as a mean of individual questions with a final score range of 0 to 10 cm; 0=best and 10=worst.
Time Frame: Week 16
Population: FAS included all participants who were randomized in the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 103 | 105
Percentage of Participants | 14.6 | 41.0

3. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score at Week 16
Description: The BASFI is a participant's self-assessment of physical function represented as a mean of 10 questions, each question rated on VAS 0 to 10 cm (VAS 0 to 10 cm; 0=easy to 10=impossible), 8 of which relate to the participant's functional anatomy and 2 of which relate to a participant's ability to cope with everyday life.
Time Frame: Baseline and Week 16
Population: FAS included all participants who were randomized in the study. Here, 'N' (Number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 98 | 105
Units on a Scale | -0.471 (1.9558) | -2.386 (2.1300)

4. Primary Outcome: Percentage of Participants Who Achieved at Least 20 Percent Improvement From Baseline in the Assessment of SpondyloArthritis International Society (ASAS 20) at Week 16
Description: ASAS 20 defined as 20 percent (%) improvement compared to baseline in the ASAS Working Group criteria: that is, greater than or equal to (>=)20% improvement from baseline in at least 3 of the 4 domains: patient's global assessment of disease activity (0=very well,10 =very poor), total back pain (0=no pain,10=most severe pain), function (self-assessment using BASFI [0=no functional impairment to 10= maximal impairment]), inflammation (0=none,10=very severe) with an absolute improvement of at least 1 (0-10 centimeter (cm) visual analogue scale [VAS]), and an absence of deterioration (defined as >=20% worsening and absolute worsening of at least 1 on a 0-10 cm scale) in the potential remaining domain.
Time Frame: Week 16
Population: The full analysis set (FAS) included all participants who were randomized in the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 103 | 105
Percentage of Participants | 26.2 | 73.3
Statistical Analysis 1: Comparison: Group 1: Placebo Then Golimumab vs Group 2: Golimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in Percentage = 47.1, 95% CI 2-sided [35.18 to 58.99]

5. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 16
Description: The Medical Outcome Study health measure SF-36 questionnaire is a well-validated and widely used quality-of-life instrument. It is a self-administered survey that consists of 8 multi-item scales: The 4 subscales of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and the 4 subscales of the SF-36 comprises the MCS score (vitality, social functioning, role-emotional, and mental health). PCS and MCS are scored from 0 to 100 with higher scores indicating better health (worst value is 0 and best value is 100), which are scored using a norm-based system where linear transformations are performed to transform scores to a mean of 50 and standard deviation of 10.
Time Frame: Baseline and Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 98 | 104
Units on a Scale | 2.86 (6.177) | 8.52 (7.535)

6. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36) Mental Component Summary (MCS) Score at Week 16
Description: The Medical Outcome Study health measure SF-36 questionnaire is a well-validated and widely used quality-of-life instrument. It is a self-administered survey that consists of 8 multi-item scales: The 4 subscales of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and the 4 subscales of the SF-36 comprises the MCS score(vitality, social functioning, role-emotional, and mental health). PCS and MCS are scored from 0 to 100 with higher scores indicating better health (worst value is 0 and best value is 100), which are scored using a norm-based system where linear transformations are performed to transform scores to a mean of 50 and standard deviation of 10.
Time Frame: Baseline and Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 98 | 104
Units on a Scale | 0.78 (10.004) | 6.47 (9.122)

7. Secondary Outcome: Percentage of Participants With Low Level of Disease Activity (ASAS Partial Remission) at Week 16
Description: Low level of disease activity was measured by criteria for ASAS partial remission, defined as a value below 2 on a scale of 0 to 10 cm in each of the 4 ASAS domains: patient's global assessment of disease activity, total back pain, function (BASFI), inflammation.
Time Frame: Week 16
Population: FAS included all participants who were randomized in the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 103 | 105
Percentage of Participants | 3.9 | 16.2

8. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 16
Description: The ASQoL is a self-administered health-related quality of life (HRQOL) instrument. It consists of 18 items requesting a Yes or No response to questions related to the impact of the disease/condition (including pain) on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. A score of 1 is given to a response of "yes" on each item and all item scores are summed to a total score with a range of 0 to 18. Higher scores indicate worse HRQOL.
Time Frame: Baseline and Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 98 | 104
Units on Scale | -1.8 (4.57) | -5.4 (5.01)

9. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 16
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: tragus to wall distance, lumbar flexion, cervical rotation, lumbar side flexion, and intermalleolar distance. Each measure was scored 0-2 (0=normal mobility/mild disease involvement, 1=moderate disease involvement, 2=severe disease involvement) to give a final total BASMI score ranging from 0 to 10. The higher the BASMI score, the more severe was the participant's limitation of movement due to their AS.
Time Frame: Baseline and Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Group 1: Placebo Then Golimumab | Group 2: Golimumab
Number analyzed (Participants) | 96 | 100
Units on Scale | -0.15 (0.737) | -0.73 (0.910)

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Description: Safety Analysis set included all participants who received at least 1 dose of study drug. Participants who received placebo and crossed over to golimumab were included in placebo then golimumab 2 mg/kg arm and who received at least 1 dose of golimumab were included in placebo then golimumab 2 mg/kg and golimumab 2 mg/kg arms for safety analysis.
Groups:
- Placebo: Participants who received placebo only (at least 1 dose) through Week 16. Follow-up was based on the period the participant was receiving placebo (from Week 0) up to the first golimumab 2 mg/kg dose for this treatment group.
- Placebo Then Golimumab 2 mg/kg: Participants who received placebo were crossed over to golimumab 2 mg/kg at Week 16. Participants may have also inadvertently received golimumab 2 mg/kg prior to Week 16. Participants may have missed one or more golimumab doses. Follow-up started from the first golimumab 2 mg/kg dose for this treatment group. Participants who inadvertently received golimumab 2 mg/kg prior to Week 16 were applicable to include in this group.
- Golimumab 2 mg/kg: Participants who received at least one dose of 2 mg/kg golimumab from Week 0 onward. Follow-up started from the first golimumab 2 mg/kg dose for this treatment group.
Arm/Group | Placebo | Placebo Then Golimumab 2 mg/kg | Golimumab 2 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/103 | 1/99 | 6/105
Other Adverse Events (participants affected / at risk) | 3/103 | 16/99 | 32/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=103) | Placebo Then Golimumab 2 mg/kg (N=99) | Golimumab 2 mg/kg (N=105)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=103) | Placebo Then Golimumab 2 mg/kg (N=99) | Golimumab 2 mg/kg (N=105)
Nasopharyngitis (Infections and infestations) | 1 | 7 | 17
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 12
Alanine aminotransferase increased (Investigations) | 0 | 5 | 7
Headache (Nervous system disorders) | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.